CLINICAL TRIAL: NCT06548893
Title: Group-based Acceptance and Commitment Therapy for Obsessive Compulsive Disorder: A Clinical Trial
Brief Title: Acceptance and Commitment Therapy (ACT) in Groups for Obsessive Compulsive Disorder: A Clinical Trial in Brazil
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Paraná (Other)
Responsible Party: Principal Investigator, Luciana Midori Samezima, Ms, Universidade Federal do Paraná
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 61795622.3.0000.0096
Record Dates: First submitted 2024-08-08; First posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: OCD; Obsessive-compulsive disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Psychotherapy, Group; Acceptance and Commitment Therapy; Psychotherapy

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Only the team member who will apply the questionnaires/scales will be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group psychotherapy with ACT (Experimental): 16 sessions of group psychotherapy based on ACT + exposure with response prevention (EPR)
  Interventions: Other: Group acceptance and commitment therapy (ACT)
- Treatment as usual (No Intervention): Patients will follow their usual treatment, without adding ACT-based group psychotherapy

INTERVENTIONS:
Other: Group acceptance and commitment therapy (ACT) — Group psychotherapy based on ACT + EPR
  Other Names: Group Psychotherapy; Acceptance and Commitment Therapy; Psychotherapy
  Arms: Group psychotherapy with ACT

SUMMARY:
The goal of this clinical trial is to learn if Acceptance and Commitment Therapy (ACT) + Exposure and Response Prevention (ERP) in Group is effective to Obsessive Compulsive Disorder (OCD) in adults.

Researchers will compare intervention to control group to see if those who attend the group therapy have better results than control group.

Participants will go through a 16-week group therapy based on a protocol designed by Michael Twohig (Twohig et al, 2018).

* Participants will not have any medication adjustment during therapy
* Participants will be assessed 3 times throughout the therapy, plus an assessment in a 6-month follow-up.

DETAILED DESCRIPTION:
The goal of this clinical trial is to learn if Acceptance and Commitment Therapy (ACT) + Exposure and Response Prevention (ERP) in Group is effective to Obsessive Compulsive Disorder (OCD) in adults. The main questions it aims to answer are:

* Can ACT in groups help decrease the severity of OCD symptoms?
* Can ACT in groups help increase psychological flexibility in this group?
* Can ACT in groups help increase quality of life in this group?

Researchers will compare intervention (n=16) to control group (n=8) to see if those who attend the group therapy have better results than control group.

We will perform an unequal randomization in a 2:1 ratio, in blocks of 6, for allocation to each group. The assessor of the outcomes of interest will be blinded to the group to which the participant was assigned

Participants will go through a 16-week group therapy based on a protocol designed by Michael Twohig (Twohig et al, 2018).

* Participants will not have any medication adjustment during therapy
* Participants will be assessed 3 times throughout the therapy, plus an assessment in a 6-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* OCD diagnosis according to DMS-5/ Minimum score of 20 in YBOCS

Exclusion Criteria:

* Psychotic disorder, maniac episode, intellectual disability, Chemical dependency, Suicidal risk, another current psychotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-08-10 (Actual); Primary Completion 2025-06-20 (Estimated); Study Completion 2026-06-20 (Estimated)

PRIMARY OUTCOMES:
Yale-Brown Obsessive-Compulsive Scale (YBOCS) | 10 months (4-month intervention + 6-month follow-up)
  Measure for assessing the presence and severity of obsessive-compulsive disorder (OCD) symptoms.

SECONDARY OUTCOMES:
Acceptance and Commitment Therapy Processes (CompACT) | 10 months (4-month intervention + 6-month follow-up)
  Measure of psychological flexibility
Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-SV) | 10 months (4-month intervention + 6-month follow-up)
  Measures of the degree of enjoyment and satisfaction experienced by subjects in various areas of dally functioning
Depression Anxiety and Stress Scale (DASS) | 10 months (4-month intervention + 6-month follow-up)
  Set of self-report scales designed to measure the emotional states of depression, anxiety and stress.
AAQ for Obsessions and Compulsions (AAQ-OC) | 10 months (4-month intervention + 6-month follow-up)
  Self-report measure of experiential avoidance in response to unwanted intrusive thoughts.
Affective Style Questionnaire (ASQ) | 10 months (4-month intervention + 6-month follow-up)
  Brief instrument to measure individual differences in emotion regulation
Clinical Global Impressions (CGI) Scale, | 10 months (4-month intervention + 6-month follow-up)
  Quantify and track patient progress and treatment response over time.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriela M Ferreira, MD, PhD, Principal Investigator — Universidade Federal do Paraná
Locations (1):
- Universidade Federal Do Paraná, Curitiba, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Twohig MP, Abramowitz JS, Smith BM, Fabricant LE, Jacoby RJ, Morrison KL, Bluett EJ, Reuman L, Blakey SM, Ledermann T. Adding acceptance and commitment therapy to exposure and response prevention for obsessive-compulsive disorder: A randomized controlled trial. Behav Res Ther. 2018 Sep;108:1-9. doi: 10.1016/j.brat.2018.06.005. Epub 2018 Jun 22. PMID 29966992
- See also: ACT+ERP for OCD: This is a 16-session twice-weekly therapist manual for OCD describing ERP conducted from an ACT framework. — https://www.utahact.com/treatment-protocols.html